CLINICAL TRIAL: NCT01919437
Title: Comparison of Methamphetamine-Dependent and Healthy Volunteers Using a Web-Enabled Cognitive Neuropsychological Evaluation System
Acronym: 5I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: Creare, Inc. (Industry)
Responsible Party: Principal Investigator, John Mendelson, MD, Senior Scientist, California Pacific Medical Center Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011.118-2
Record Dates: First submitted 2013-05-29; First posted 2013-08-09 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Methamphetamine Dependence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Web-Enabled Cognitive Neuropsychological Evaluation System (Experimental)
  Interventions: Device: Web-Enabled Cognitive Neuropsychological Evaluation System

INTERVENTIONS:
Device: Web-Enabled Cognitive Neuropsychological Evaluation System

SUMMARY:
The purpose of this study is to develop the technology infrastructure for a mobile Web-based cognitive and neuropsychological assessment of substance abusers, and to perform a pilot trial using neurocognitive tasks designed to demonstrate that our system is statistically comparable to current clinical practice.

The primary hypotheses are that results collected using a web-based data collection platform will be comparable (but not necessarily equivalent) to data collected under controlled laboratory conditions, that methamphetamine (MA) dependent participants will have worsened neurocognitive performance compared to healthy volunteers, and the platform will be acceptable to participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 55.
* Ability to give informed consent.

Exclusion Criteria:

* Unwilling or unable to access the web over a cell phone or living in an area with no cell phone service.
* Any medical, psychiatric, or other condition that, in the opinion of the investigator, would preclude safe, consistent, or useful participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of neurocognitive task results | 2 weeks
  Results collected using a web-based data collection platform will be comparable (but not necessarily equivalent) to data collected under controlled laboratory conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- CPMC Addiction & Pharmacology Research Laboratory, San Francisco, California, United States